CLINICAL TRIAL: NCT07316634
Title: Correlation Between Postoperative Blood Pressure Variability, Perfusion Index and Perioperative Adverse Events in Cardiac Surgery: A Single-Center Prospective Observational Cohort Study
Brief Title: Correlation Between Postoperative Blood Pressure Variability, Perfusion Index and Perioperative Adverse Events in Cardiac Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Nan Liu, head of department, Beijing Anzhen Hospital
Other Study IDs: KS2025145
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Surgery Intensive Care Treatment; Hemodynamics
Keywords: Blood Pressure Variability; Perfusion Index; Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult Patients After Cardiac Surgery
  Interventions: Other: Blood Pressure Variability and Perfusion Index

INTERVENTIONS:
Other: Blood Pressure Variability and Perfusion Index — All patients in this cohort will undergo invasive hemodynamic monitoring and noninvasive pulse oximetry, postoperative 24-hour blood pressure variability (from minute-to-minute invasive arterial pressure data) and perfusion index (from half-hourly recordings) were obtained through these monitoring modalities.

SUMMARY:
In patients after cardiac surgery, disturbances in macrocirculatory fluctuations and tissue perfusion commonly coexist. The stress state induced by factors such as surgical manipulation, cardiopulmonary bypass, anesthetic agents, pain, and ischemia-reperfusion injury, along with the use of vasoactive drugs postoperatively, often leads to increased blood pressure fluctuations in the early postoperative period. Additionally, dysregulation of organ blood flow autoregulation post-surgery contributes to peripheral circulatory impairment, rendering perfusion pressure an unreliable indicator of actual organ perfusion. We aim to assess postoperative blood pressure fluctuation using blood pressure variability and evaluate peripheral circulatory status via the perfusion index. In this prospective cohort study, we will examine the correlation between these two parameters and perioperative adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age at surgery ≥ 18 years

  * Patients admitted to the ICU for the first time after undergoing their first cardiac surgical procedure during the current hospitalization ③ Expected to receive continuous invasive blood pressure monitoring and noninvasive pulse oximetry monitoring for at least 12 hours postoperatively in the ICU ④ Written or verbal informed consent obtained from the patient or their family members

Exclusion Criteria:

* Patients with severe peripheral vascular disease in the arm used for noninvasive pulse oximetry monitoring

  * Patients not undergoing invasive hemodynamic monitoring ③ Patients requiring preoperative or intraoperative support with IABP or ECMO

    * Patients expected to have incomplete postoperative monitoring data or a monitoring duration of less than 12 hours

      * Postoperative patients who are not admitted to the ICU for the first time during the current hospitalization ⑥ Patients admitted to the ICU prior to undergoing cardiac surgery ⑦ Patients with critically insufficient baseline preoperative data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery at Beijing Anzhen Hospital, Capital Medical University
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of the composite endpoint of adverse events within 30 days postoperatively | Within 30 days after surgery
  Total incidence of death, stroke, perioperative myocardial infarction, infection, reoperation, and continuous renal replacement therapy.
  Diagnostic criteria:
  Stroke was characterized by a new focal deficit associated with a compatible image on computed tomography.
  Perioperative myocardial infarction was diagnosed when cardiac troponin I shows an acute change with at least one value exceeding the 99th percentile upper reference limit, along with one of the following: new pathologic Q waves, imaging evidence of coronary artery occlusion, or imaging evidence of new loss of viable myocardium.
  Infection was considered if one of the following diagnoses was made by an Infectious Disease specialist who followed specific protocols: 1) Pneumonia; 2) Catheter related blood stream infection; 3) Sternal wound infection or osteomyelitis.

SECONDARY OUTCOMES:
Incidence of low cardiac output syndrome within 30 days postoperatively. | Within 30 days after surgery
  Diagnostic criteria: Cardiac index < 2.0 L/min/m².
Incidence of acute kidney injury within 30 days postoperatively. | Within 30 days after surgery
  Diagnostic criteria are based on the KDIGO guidelines.
Incidence of acute respiratory distress syndrome within 30 days postoperatively | Within 30 days after surgery
  Diagnostic criteria are based on the 2012 Berlin definition of ARDS.
Incidence of new-onset atrial arrhythmias within 30 days postoperatively. | Within 30 days after surgery
  Diagnostic criteria: atrial fibrillation or atrial flutter lasting more than 1 hour on continuous electrocardiographic monitoring, requiring pharmacological or electrical cardioversion.
Incidence of prolonged ventilation (>24 hours) within 30 days postoperatively. | Within 30 days after surgery
Length of intensive care unit stay | Within 30 days after surgery

IPD SHARING:
Plan to Share IPD: Undecided